CLINICAL TRIAL: NCT02751333
Title: Esophageal Stent Migration With Endoscopic Suture Fixation Compared to Standard Deployment in the Management of Benign Esophageal Pathology: A Randomized Controlled Trial
Brief Title: Esophageal Stent Migration With Endoscopic Suture Fixation Compared to Standard Deployment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The reason was the fact that the study was not clinically feasible.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Mouen Khashab, Associate professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00091684
Record Dates: First submitted 2016-04-18; First posted 2016-04-26 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Esophageal Strictures; Esophageal Leak; Esophageal Perforation; Esophageal Fistula; Endostitch; Esophageal Stent
Keywords: Esophageal stricture; Esophageal leak; Esophageal perforation; Esophageal fistula; Endostitch; Esophageal stent
MeSH Terms: conditions — Esophageal Stenosis; Esophageal Perforation; Esophageal Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FCSEMS with Endostitching (ES) (Active Comparator): General anesthesia or conscious sedation will be started and an upper endoscope will be inserted into the participants mouth and advanced into the stomach. Endoscopic stenting with a fully covered self-expanding metal stents (FCSEMS) will then be performed. Once the stent is in place, the endoscope will be withdrawn from the participant to set-up the endostitch device unto the endoscope. Bites are taken separately with the first on the esophageal mucosa followed by a second on the stent itself and finishing with a last bite on esophageal mucosa. A cinch is then used to secure the deployed suture. An attempt at placing 2 sutures will be performed. Stent removal will then be performed at 8-weeks post-stent insertion.
  Interventions: Procedure: FCSEMS with Endostitch (ES); Device: Fully Covered Self-Expanding Metal Stents (FCSEMS); Device: EndoStitch (ES) with the OverStitchTM system
- FCSEMS with No Suturing (NS) (Active Comparator): The procedure will be done in the same manner with same endoscopic technique, stent deployment, and timing of stent removal. The only difference would be the lack of suturing and naturally the need for suture cutting at stent removal.
  Interventions: Procedure: FCSEMS with No Suturing (NS); Device: Fully Covered Self-Expanding Metal Stents (FCSEMS)

INTERVENTIONS:
Procedure: FCSEMS with Endostitch (ES) — The fixation of FCSEMS using endostitch (ES) with the OverStitchTM system to prevent migration.
  Arms: FCSEMS with Endostitching (ES)
Procedure: FCSEMS with No Suturing (NS) — The insertion of FCSEMS with no suturing.
  Arms: FCSEMS with No Suturing (NS)
Device: Fully Covered Self-Expanding Metal Stents (FCSEMS) — This is the stent that will be used to treat the esophageal pathology in both groups
Device: EndoStitch (ES) with the OverStitchTM system — This is the device used to apply the stitches to the stent in participants randomized to stent suturing.
  Arms: FCSEMS with Endostitching (ES)

SUMMARY:
Esophageal stents are commonly used for benign esophageal pathology, especially strictures or esophageal mucosal defects such as leaks, fistulae, or perforations. The major limiting factor to stent placement is the high migration rate of the stent. Investigators are trying to prospectively evaluate the efficacy of endostitch in preventing stent migration in benign esophageal disease in comparison with standard, fully covered self-expanding metal stents (FCSEMS) placement without fixation.

DETAILED DESCRIPTION:
The use of removable, fully covered self-expanding metal stents (FCSEMS) in the management of benign esophageal pathology has been increasingly applied in recent years. Several studies have shown promising results with its application in esophageal perforation, fistula, or leak, and refractory benign strictures. However, the major limiting factor to successful treatment with FCSEMS in this setting is the substantial migration rates.

Different strategies has been used to secure esophageal stents but to little success. Several tertiary institutions including investigators have adopted the use of endostitch (ES) with the OverStitchTM system (Apollo Endosurgery, Austin, Texas) as the preferred method for stent fixation. Animal ex-vivo studies have confirmed the greater anchoring ability and tensile strength with this method when compared to esophageal stenting alone or with through the endoscope clip fixation while retrospective series have shown promising results with lower rates of stent migration when compared to conventional stent insertion. However, although the use of endostitch stent fixation has been used in several centers in the United-States with strong retrospective data (including investigators data), no prospective randomized controlled trial have confirmed its effectiveness in preventing stent migration.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age 18 years and older
2. Patients with esophageal refractory benign strictures (peptic, anastomotic, caustic, radiation, and idiopathic) where a 14 mm luminal diameter cannot be achieved over 2 dilation sessions at 1-3-week intervals.
3. Patients with esophageal leak, perforation, or fistula referred for endoscopic stenting
4. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Pediatric patients age under 18 years
2. Pregnant or breastfeeding patients
3. Patients with malignant esophageal lesions, primary or metastatic, requiring endoscopic stenting (all females of child bearing age will undergo urine pregnancy testing as per standard1 preprocedural testing)
4. Benign strictures not having had two attempts at endoscopic dilation
5. Uncorrectable coagulopathy defined by partial thromboplastin time (PTT) greater than 50 sec, or international normalized ratio (INR) greater than 1.5
6. Uncorrectable thrombocytopenia with platelet count less than 50, 000

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Stent Migration as assessed by Symptoms suggestive of stent migration or objective evidence of migration on radiological imaging or endoscopy. | Up to 6 months
  Subjects returning to the hospital following stent placement with symptoms suggestive of stent migration such as fever, abdominal or chest pain, nausea/vomiting, and dysphagia with objective evidence of stent migration either on radiological imaging or endoscopy.

SECONDARY OUTCOMES:
Clinical success of stent deployment as assessed by the relief of the pre-stent dysphagia | 4 weeks, 6 months post-stent removal
  Dysphagia relief as assessed by the validated dysphagia score
Procedure time | During procedure
  Time required for stent placement with/without endostitch
Stent insertion complication rate | 3 days post-stent insertion, 4 weeks post-stent removal
  All complications related to stent insertion other than stent migration will be recorded with a preset questionnaire to measure the frequency of complications related to stent insertion.
Quality of life | prior to stent insertion and 6 months post-stent removal
  Quality of life as measured by the SF-36 (Short Form health survey) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mouen Khashab, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States